CLINICAL TRIAL: NCT00691015
Title: A Phase II Study of Sirolimus, Tacrolimus and Thymoglobulin®, as Graft-versus-Host- Disease Prophylaxis in Patients Undergoing Unrelated Donor Hematopoietic Cell Transplantation
Brief Title: Sirolimus, Tacrolimus, and Antithymocyte Globulin in Preventing Graft-Versus-Host Disease in Patients With Hematologic Cancer Who Are Undergoing Donor Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Zaid Al-Kadhimi, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007-127; P30CA022453 (NIH); GENZ-WSU-2007-127; 2007-127 (Other: Barbara Ann Karmanos Cancer Institute)
Record Dates: First submitted 2008-06-04; First posted 2008-06-05 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-05

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); chronic phase chronic myelogenous leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; secondary acute myeloid leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; de novo myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; primary myelofibrosis; atypical chronic myeloid leukemia, BCR-ABL negative; chronic eosinophilic leukemia; chronic myelomonocytic leukemia; chronic neutrophilic leukemia
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Acute; Primary Myelofibrosis; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic | interventions — Rituximab; Busulfan; Carmustine; carmustine, poliferprosan 20 drug combination; Cyclophosphamide; Cytarabine; Etoposide; etoposide phosphate; fludarabine phosphate; Melphalan; Whole-Body Irradiation; Radiotherapy; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy or chemotherapy + total body irradiation (Experimental): Standard of care (SOC) chemotherapy or ( SOC) chemotherapy + total body irradiation (TBI) of one of the following regimens:
  Regimen I: Patients receive fludarabine phosphate IV and busulfan IV; anti-thymocyte globulin IV.
  Regimen II: Patients undergo total body irradiation (TBI) twice daily for 8 fractions and receive etoposide IV;anti-thymocyte globulin IV.
  Regimen III: Patients undergo TBI once or twice daily for 11 fractions and receive cyclophosphamide IV; anti-thymocyte globulin IV.
  Regimen IV: Patients undergo TBI and receive fludarabine phosphate IV and busulfan IV; anti-thymocyte globulin IV.
  Regimen V: Patients receive carmustine IV, etoposide IV, cytarabine IV, and melphalan IV. Some patients also receive rituximab IV; anti-thymocyte globulin IV.
  Regimen VI: Patients receive fludarabine phosphate IV and melphalan IV. Some patients also undergo TBI; anti-thymocyte globulin IV.
  Interventions: Biological: rituximab; Drug: busulfan; Drug: carmustine; Drug: cyclophosphamide; Drug: cytarabine; Drug: etoposide; Drug: fludarabine phosphate; Drug: melphalan; Radiation: total body irradiation (TBI); Drug: anti-thymocyte globulin IV

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: Rituxan; MabThera; Zytux
Drug: busulfan — Given IV
  Other Names: Busulfex; Myleran
Drug: carmustine — Given IV
  Other Names: Bicnu; Gliadel
Drug: cyclophosphamide — Given IV
  Other Names: Cytoxan; Cytoxan Lyophilized; Neosar
Drug: cytarabine — Given IV
  Other Names: Depocyt
Drug: etoposide — Given IV
  Other Names: Etopophos; Toposar
Drug: fludarabine phosphate — Given IV
  Other Names: Fludara®
Drug: melphalan — Given IV
  Other Names: Alkeran
Radiation: total body irradiation (TBI) — Given once or twice daily
  Other Names: radiotherapy
Drug: anti-thymocyte globulin IV — Given IV
  Other Names: Thymoglobulin

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, monoclonal antibodies, and radiation therapy before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving tacrolimus, sirolimus, and antithymocyte globulin before and after transplant may stop this from happening.

PURPOSE: This phase II trial is studying the side effects of giving sirolimus together with tacrolimus and antithymocyte globulin and to see how well it works in preventing graft-versus-host disease in patients with hematologic cancer who are undergoing donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the incidence and severity of acute graft-versus-host disease (GVHD) after HLA-matched or -mismatched unrelated donor peripheral blood stem cell transplantation (PBSCT) in patients with hematologic malignancies treated with immunosuppressive therapy comprising sirolimus, tacrolimus, and anti-thymocyte globulin as GVHD prophylaxis.
* To determine the safety of this regimen in these patients at 6 months after PBSCT.

Secondary

* To determine the time to engraftment (i.e., platelet and absolute neutrophil recovery) in patients treated with this regimen.
* To determine the length of hospital stay of these patients within 100 days after PBSCT.
* To determine the incidence of infections, including CMV and EBV reactivation and post-transplant lymphoproliferative disorders, in patients treated with this regimen.
* To determine the incidence of thrombotic microangiopathy and veno-occlusive disease in patients treated with this regimen.
* To determine the incidence of chronic GVHD in patients treated with this regimen.
* To determine the overall and disease-free survival of these patients at 2 years after PBSCT.
* To determine the Karnofsky performance status of these patients at baseline and at various time points after PBSCT.
* To conduct immunocorrelative studies prior to and at various time points after PBSCT.

OUTLINE:

* Conditioning regimen: Patients receive 1 of 6 conditioning regimens (standard of care treatment) between days -9 and -3, based on diagnosis and the treating physician's preference regarding regimen intensity.

  * Regimen I: Patients receive fludarabine phosphate IV and busulfan IV.
  * Regimen II: Patients undergo total body irradiation (TBI) twice daily for 8 fractions and receive etoposide IV.
  * Regimen III: Patients undergo TBI once or twice daily for 11 fractions and receive cyclophosphamide IV.
  * Regimen IV: Patients undergo TBI and receive fludarabine phosphate IV and busulfan IV.
  * Regimen V: Patients receive carmustine IV, etoposide IV, cytarabine IV, and melphalan IV. Some patients also receive rituximab IV.
  * Regimen VI: Patients receive fludarabine phosphate IV and melphalan IV. Some patients also undergo TBI.
* Allogeneic peripheral blood stem cell transplantation: Patients undergo filgrastim (G-CSF)-mobilized allogeneic peripheral blood stem cell transplantation on day 0.
* Graft-versus-host disease prophylaxis (GVHD): Patients receive tacrolimus IV continuously over 24 hours or orally and sirolimus orally beginning on day -3 and continuing until day 30 or day 90, followed by a taper in the absence of GVHD. Patients also receive anti-thymocyte globulin IV over 4-8 hours on days -3 to -1.

Blood samples are obtained at baseline and periodically during study for correlative biomarker studies. Samples are analyzed by T-cell immunophenotyping, absolute subset number quantification, and multi-parameter flow cytometry for evaluation of immune reconstitution, T-cell differentiation status, NK-cell recovery, allo-reactivity of donor T-cells after transplantation, and regulatory T-cell reconstitution.

After completion of study therapy, patients are followed periodically for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a hematological malignancy, including any of the following:

  * Non-Hodgkin lymphoma in complete remission (CR) or partial remission (PR)
  * Hodgkin lymphoma in CR or PR
  * Acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL) meeting either of the following criteria:

    * In CR
    * Not in CR and meets the following criteria:

      * Bone marrow blast < 20% within 4 weeks of transplantation
      * Peripheral blood absolute blast count < 500 per microliter on the day of initiating conditioning therapy
  * Myelodysplastic syndromes, treated or untreated
  * Chronic myeloid leukemia in chronic phase or accelerated phase
  * Multiple myeloma in CR or PR
  * Chronic lymphocytic leukemia in second or greater CR or PR
  * Myelofibrosis or other myeloproliferative disorders meeting the following criteria:

    * Bone marrow blasts < 20% within 4 weeks of transplantation
    * Peripheral blood absolute blast count < 500 per microliter on the day of initiating conditioning therapy
    * Patients with ascites not allowed
* No prior bone marrow or ex vivo engineered or processed graft (i.e., CD34+ enrichment, T-cell depletion, etc)
* Scheduled to undergo peripheral blood stem cell transplantation from a suitable HLA-matched or -mismatched unrelated donor, as determined by treating physician

  * High resolution molecular HLA typing is required for HLA class I and II
  * No more than one antigen or allele mismatch
* No documented uncontrolled CNS disease

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2
* Karnofsky PS 60-100%
* Creatinine clearance > 50 mL/min
* Bilirubin < 3 times upper limit of normal (ULN)
* ALT and AST < 3 times ULN
* LVEF > 50%
* FVC, FEV_1, or DLCO > 50% predicted

  * Patients on home oxygen not allowed
* Able to cooperate with oral medication intake
* HIV negative
* No active hepatitis B or hepatitis C
* No known contraindication to sirolimus, tacrolimus, or anti-thymocyte globulin

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zaid Al-Kadhimi, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Conditioning Regimen: Chemotherapy or chemotherapy + total body irradiation
  Standard of care (SOC) chemotherapy or ( SOC) chemotherapy + total body irradiation (TBI) of one of the following regimens:
  Regimen I: Patients receive fludarabine phosphate IV and busulfan IV.
  Regimen II: Patients undergo total body irradiation (TBI) twice daily for 8 fractions and receive etoposide IV.
  Regimen III: Patients undergo TBI once or twice daily for 11 fractions and receive cyclophosphamide IV.
  Regimen IV: Patients undergo TBI and receive fludarabine phosphate IV and busulfan IV.
  Regimen V: Patients receive carmustine IV, etoposide IV, cytarabine IV, and melphalan IV. Some patients also receive rituximab IV.
  Regimen VI: Patients receive fludarabine phosphate IV and melphalan IV. Some patients also undergo TBI.
Period: Overall Study
Arm/Group | Conditioning Regimen
Started | 48
Completed | 47
Not Completed | 1
Not completed — Refused further treatment | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All regimens were analyzed together.
  Standard of Care (SOC) Chemotherapy or Standard of Care (SOC) Chemotherapy + total body irradiation
  SOC chemotherapy or SOC chemotherapy + total body irradiation (TBI) of one of the following regimens:
  Regimen I: Patients receive fludarabine phosphate IV and busulfan IV.
  Regimen II: Patients undergo total body irradiation (TBI) twice daily for 8 fractions and receive etoposide IV.
  Regimen III: Patients undergo TBI once or twice daily for 11 fractions and receive cyclophosphamide IV.
  Regimen IV: Patients undergo TBI and receive fludarabine phosphate IV and busulfan IV.
  Regimen V: Patients receive carmustine IV, etoposide IV, cytarabine IV, and melphalan IV. Some patients also receive rituximab IV.
  Regimen VI: Patients receive fludarabine phosphate IV and melphalan IV. Some patients also undergo TBI.
Arm/Group | All Participants
Number analyzed (Participants) | 47
Age, Continuous [Median (Full Range); unit: years] | 53 [20 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 30
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Acute Graft-versus-host Disease (GVHD)
Time Frame: Within 100 days after donor peripheral blood stem cell transplantation (PBSCT) as assessed by Glucksberg criteria
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- All Participants: All regimens were analyzed together.
Arm/Group | All Participants
Number analyzed (Participants) | 47
percentage of participants | 44.7 [33.4 to 56.6]

2. Primary Outcome: Severity of Acute Graft-versus-host Disease (GVHD)
Time Frame: Within 100 days after donor peripheral blood stem cell transplantation (PBSCT) as assessed by Glucksberg criteria
Population: The patients that contracted sever acute graph versus host disease (aGVHD) from those who developed aGVHD
Measure: Number (90% Confidence Interval); unit: % of participants with severe aGVHD
Arm/Group | All Participants
Number analyzed (Participants) | 21
% of participants with severe aGVHD | 33.3 [19.2 to 51.3]

3. Primary Outcome: Safety, as Defined by Serious Adverse Events and Adverse Events Related to Study Treatment.
Time Frame: Within 6 months after PBSCT
Population: All participants
Measure: Number (95% Confidence Interval); unit: % of participants with a reported SAE
Arm/Group | All Participants
Number analyzed (Participants) | 47
% of participants with a reported SAE | 93.62 [82.46 to 98.66]

4. Secondary Outcome: Incidence of Chronic GVHD.
Time Frame: Within 2 years after PBSCT
Population: All participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 47
percentage of participants | 44.68 [30.17 to 59.88]

5. Secondary Outcome: Time to Engraftment (i.e., Absolute Neutrophil Recovery [ANC > 500/mm³] )
Time Frame: post transplant, up to 4 weeks
Population: All participants
Measure: Median (Full Range); unit: Days
Arm/Group | All Participants
Number analyzed (Participants) | 47
Days | 11 [9 to 15]

6. Secondary Outcome: Overall Survival.
Time Frame: At 2 years after PBSCT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 47
percentage of participants | 57.4 [44.9 to 73.5]

7. Secondary Outcome: Incidence of Infections, Including Bacterial, Fungal, and Viral Infections (i.e., CMV and EBV Reactivation, Including Post-transplant Lymphoproliferative Disorders)
Time Frame: Within 6 months after PBSCT
Population: All participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 47
percentage of participants | 80.85 [66.74 to 90.85]

8. Secondary Outcome: Karnofsky Performance Status Performance Status
Description: 100 - Normal; no complaints; no evidence of disease. 90 - Able to carry on normal activity; minor signs or symptoms of disease. 80 - Normal activity with effort; some signs or symptoms of disease. 70 - Cares for self; unable to carry on normal activity or to do active work. 60 - Requires occasional assistance, but is able to care for most of their personal needs.
  50 - Requires considerable assistance and frequent medical care. 40 - Disabled; requires special care and assistance. 30 - Severely disabled; hospital admission is indicated although death not imminent.
  20 - Very sick; hospital admission necessary; active supportive treatment necessary.
  10 - Moribund; fatal processes progressing rapidly. 0 - Dead
Time Frame: At 90 days after PBSCT
Population: All participants
Measure: Median (Full Range); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 47
units on a scale | 80 [60 to 100]

ADVERSE EVENTS:
Arm/Group | Conditioning Regimen
Serious Adverse Events (participants affected / at risk) | 44/47
Other Adverse Events (participants affected / at risk) | 0/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conditioning Regimen (N=47)
alanine aminotransferase (ALT) increased (Investigations) | 6 (6)
alanine aminotransferase (ALT), SGPT (Investigations) | 2 (2)
aspartate aminotransferase (AST) increased (Investigations) | 7 (7)
aspartate aminotransferase (AST) increased, SGOT (Investigations) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 4 (4)
Acute Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alkaline Phosphatase increased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 4 (4)
Bilirubin increased (Investigations) | 9 (9)
Blood/Bone Marrow (Blood and lymphatic system disorders) | 1 (1)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1)
Calcium serum - low (Metabolism and nutrition disorders) | 6 (6)
Cardiac ischemia/infarction (Cardiac disorders) | 3 (3)
Cardiac troponin I increased (Investigations) | 3 (3)
Cardiopulmonary arrest (Cardiac disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 7 (7)
Confusion (Psychiatric disorders) | 5 (5)
Creatinine increased (Investigations) | 7 (7)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Dermatology/Skin - palmar erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Encephalopathy (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2)
Glucose (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 12 (12)
Hemoglobin (Investigations) | 11 (11)
Hemorrhage, GI (General disorders) | 4 (4)
Hemorrhage, GI-Liver (Gastrointestinal disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hemorrhage, pulmonary/upper respiratory/lung (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hemorrhage/bleeding associated with surgery, intra-operative or postoperative (Injury, poisoning and procedural complications) | 1 (1)
Hepatobiliary/Pancreas - Other (VOD/SOS) (Hepatobiliary disorders) | 3 (3)
Hypertension (Vascular disorders) | 4 (4)
Hypotension (Vascular disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Ileus (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 24 (24)
Infection BK (Infections and infestations) | 6 (6)
Infection CMV (Infections and infestations) | 6 (6)
Infection EBV (Infections and infestations) | 4 (4)
Infection HSV (Infections and infestations) | 2 (2)
Infection VZV in CSF (Infections and infestations) | 1 (1)
Infections aspergillus (Infections and infestations) | 2 (2)
Infection Pulmonary (Infections and infestations) | 1 (1)
infection, with normal ANC (Infections and infestations) | 11 (11)
Infection-Pulmonary/Upper Resp. (Infections and infestations) | 2 (2)
Iron Overload (Metabolism and nutrition disorders) | 6 (6)
Left Ventricular diastolic dysfunction (Cardiac disorders) | 1 (1)
Left Ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Leukocytes (Blood and lymphatic system disorders) | 12 (12)
Lipase (Investigations) | 2 (2)
Liver Dysfunction/Failure (Hepatobiliary disorders) | 1 (1)
Lymphocytes (Investigations) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 11 (11)
Magnesium, Serum high (Metabolism and nutrition disorders) | 2 (2)
Magnesium, Serum low (Metabolism and nutrition disorders) | 1 (1)
mood alteration (Psychiatric disorders) | 1 (1)
Mucositis/stomatis-large bowel (Gastrointestinal disorders) | 2 (2)
Mucositis/stomatis-Small bowel (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7)
Neutrophils (Investigations) | 11 (11)
Other-Right side facial droop (Nervous system disorders) | 1 (1)
Pain Pulmonary/Respiratroy-throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain-Gastrointestinal-Abdominal NOS (Gastrointestinal disorders) | 1 (1)
Pain-mid/back, hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain-Cardiovascular-cardiac/heart (Cardiac disorders) | 1 (1)
Pain-Gastrointestinal-oral cavity (Gastrointestinal disorders) | 4 (4)
Pain-gastrointestinal-stomach (Gastrointestinal disorders) | 1 (1)
Pain-Musculoskeletal-Back (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain-Musculoskeletal-Bone (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain-Neurology-head/headache (Nervous system disorders) | 2 (2)
Pain-Neurology-headache (Nervous system disorders) | 1 (1)
pain-renal/genitourinary (Renal and urinary disorders) | 1 (1)
pain-chest wall (Musculoskeletal and connective tissue disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Platelets (Investigations) | 12 (12)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Potassium, Serum high (Metabolism and nutrition disorders) | 7 (7)
Potassium, serum low (Metabolism and nutrition disorders) | 4 (4)
prolonged intubation (Investigations) | 3 (3)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 10 (10)
Renal-other-Acute Renal Failure (Renal and urinary disorders) | 5 (5)
Rigors/chills (General disorders) | 2 (2)
Sodium, Serum-low (Metabolism and nutrition disorders) | 4 (4)
Somnolence/depressed level of consciousness (Nervous system disorders) | 4 (4)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 2 (2)
Thrombosis/embolism/thrombus (Vascular disorders) | 1 (1)
Thrombosis/embolism (left lower extremity) (Vascular disorders) | 1 (1)
Thrombosis/embolism (pulmonary) (Vascular disorders) | 1 (1)
Thrombotic microangiopathy (Vascular disorders) | 4 (4)
Ventricular arrhythmia-ventricular tachycardia (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Death-disease progression (General disorders) | 2 (2)
Death-disease progression NOS (General disorders) | 1 (1)
Death-GVHD (General disorders) | 1 (1)
Death SOS (General disorders) | 1 (1)
Death-cGVHD (General disorders) | 3 (3)
Death-aGVHD/infection (General disorders) | 1 (1)
Death-Multi organ failure (General disorders) | 2 (2)
Death-Multi organ failure/SOS (General disorders) | 1 (1)
Death-Multi organ failure/Sepsis (Infections and infestations) | 2 (2)
Death-pancytopenia possible bleed (General disorders) | 1 (1)
Death-Disease progression (from 2nd BMT not associated with this protocol) (General disorders) | 1 (1)
Death-aGVHD (General disorders) | 1 (1)
Death-intersititial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No